CLINICAL TRIAL: NCT06174220
Title: Targeted Therapy With Glycogen Synthase Kinase-3 Inhibition for Arrhythmogenic Cardiomyopathy
Acronym: TaRGET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Population Health Research Institute (Other); Canadian Institutes of Health Research (CIHR) (Other Government); AMO Pharma (Unknown); Hearts in Rhythm Organization (HiRO) (Unknown); Canadian SADS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRI.TaRGET
Record Dates: First submitted 2023-12-01; First posted 2023-12-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-04

CONDITIONS: Arrhythmogenic Cardiomyopathy; Arrhythmogenic Right Ventricular Cardiomyopathy
Keywords: sudden cardiac death, ventricular cardiomyopathy, genetics, arrhythmia
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Death, Sudden, Cardiac; Arrhythmias, Cardiac | interventions — tideglusib

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio using an automated central, web-based system within 30 days of completing their baseline Holter. Randomization will be stratified by TMEM43-p.S358L variant status.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tideglusib (Active Comparator): Randomization to Tideglusib 1g po daily or matching placebo
  Interventions: Drug: Tideglusib
- Placebo (Placebo Comparator): Randomization to matching placebo 1g po daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tideglusib — Tideglusib 1g po daily
  Arms: Tideglusib
Drug: Placebo — Matching placebo 1g po daily
  Arms: Placebo

SUMMARY:
The TaRGET study is a multi-centre, prospective, randomized, double-blind, placebo-controlled trial designed to evaluate the potential therapeutic efficacy of tideglusib, a glycogen synthase kinase-3 β inhibitor, in genotype positive arrhythmogenic cardiomyopathy.

DETAILED DESCRIPTION:
Arrhythmogenic cardiomyopathy (ACM) is a heritable form of structural heart disease characterized by myocardial fibrosis that confers vulnerability to malignant ventricular arrhythmias and sudden cardiac death (SCD). A subgroup of cases preferentially involves the right ventricle and is termed arrhythmogenic right ventricular cardiomyopathy (ARVC). Although an increasingly diverse set of genes have been implicated in ACM, its most prominent genetic culprits are constituents of the desmosome, a specialized cellular structure within the intercalated disc that mediates intercellular adhesion. An additional ACM genetic subtype develops secondary to the TMEM43-p.S358L variant and is associated with an aggressive clinical phenotype, particularly among males.

Despite dramatic progress in unravelling the genetic underpinnings of ACM, insight into its pathophysiology remains modest. A lack of understanding of its operative biological pathways has rendered development of tailored treatments challenging, leading to approaches to medical therapy being largely adopted from those utilized for more common forms of cardiomyopathy. An implantable cardioverter defibrillator (ICD) is recommended for prevention of SCD for all ACM patients considered high risk for malignant ventricular arrhythmias, however does not address its underlying pathophysiology. Subsequent prevention of painful ICD shocks for ventricular tachycardia often requires interventions that may carry modest efficacy and significant risks for adverse events, including anti-arrhythmic drugs and invasive combined endo- and epicardial catheter ablation procedures.

In 2014, a high-throughput screen of a library of bioactive compounds against a zebrafish model of ACM identified a small molecule classified as a glycogen synthase kinase-3 (GSK3) inhibitor that successfully prevented and rescued the phenotype, findings that have subsequently been reproduced in a series of ACM murine models. GSK3 is an enzyme that modulates the activity of a broad spectrum of intracellular signaling pathways, including the canonical Wnt/β-catenin pathway, whose suppression has been suggested to exert an important role in ACM pathogenesis.

Tideglusib is an oral GSK3β inhibitor with an established safety profile in humans. Driven by promising findings observed for tideglusib in ACM mouse models, we now seek to evaluate its potential efficacy in a randomized clinical trial involving genotype positive ACM patients.

ELIGIBILITY:
Inclusion Criteria:

* A pathogenic or likely pathogenic desmosomal (PKP2, DSG2, DSC2, DSP, or JUP*) rare variant OR the TMEM43-p.S358L variant

  *JUP carriers must be homozygous or compound heterozygous
* Mean ≥ 500 PVCs per 24 hours on a baseline screening 7-day Holter monitor
* Clinical ACM diagnosis or recognition of genetic carrier status for ≥ 6 months prior to screening

Exclusion Criteria:

* NYHA class IV heart failure
* Ventricular scar secondary to coronary artery disease
* Initiation, cessation, or dose change of a Class I or III anti-arrhythmic drug in the 3 months prior to screening
* Any potentially harmful chronic liver disease
* ALT value > 2X the upper limit of the normal reference range at Screening
* Total bilirubin value greater than the upper limit of the normal reference range at Screening, unless documented Gilbert's syndrome. For individuals with Gilbert's syndrome, total bilirubin value greater than 2-fold the upper limit of the normal reference range at Screening.
* A history of alcohol or illicit substance use disorders
* Regular and long-term use of strong CYP3A4 inhibitors, including clarithromycin, telithromycin, ketoconazole, itraconazole, posaconazole, nefazodone, idinavir and ritonavir
* Serum creatinine > 150 micromole/L or creatinine clearance ≤ 60 mL/min (according to Cockcroft-Gault formula) at Screening
* Pregnant at time of enrollment and women of childbearing age who do not use a highly effective form of contraception
* Males, engaged in sexual relations with a female of child-bearing potential, not using an acceptable contraceptive method if not surgically sterile
* Patients unwilling to provide informed consent or comply with follow-up
* Hypersensitivity to tideglusib or any components of its formulation, including allergy to strawberry
* Concurrent use of drugs metabolized by CYP3A4 with a narrow therapeutic window e.g. warfarin and digoxin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
PVC burden | Baseline and 6 months
  Change in mean PVC count per 24 hours on 7-day Holter

SECONDARY OUTCOMES:
Ventricular strain | Baseline and 6 months
  Change in ventricular strain on echocardiography
Implantable cardioverter-defibrillator (ICD) therapies | Baseline and 6 months
  Number of ICD therapies (shock or anti-tachycardia pacing)
Sustained ventricular tachycardia (VT) events | Baseline and 6 months
  Number of sustained VT events (defined as symptomatic or duration > 30 seconds and > 100bpm)

CONTACTS AND LOCATIONS:
Overall Officials: Jason D Roberts, MD MAS, Principal Investigator — McMaster University and Population Health Research Institute
Locations (17):
- Canada (17):
  - Foothills Medical Centre, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Cardiac Arrhythmia Trials Inc., Victoria, British Columbia
  - Health Sciences Centre, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Newmarket Electrophysiologist Research Group 'NERG', Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Heart Health Institute Research Inc, Scarborough Village, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hopital du Sacré-Coeur de Montréal, Montreal, Quebec
  - University Institute of Cardiology and Pneumology of Quebec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krahn AD, Wilde AAM, Calkins H, La Gerche A, Cadrin-Tourigny J, Roberts JD, Han HC. Arrhythmogenic Right Ventricular Cardiomyopathy. JACC Clin Electrophysiol. 2022 Apr;8(4):533-553. doi: 10.1016/j.jacep.2021.12.002. PMID 35450611
- [Background] Asimaki A, Kapoor S, Plovie E, Karin Arndt A, Adams E, Liu Z, James CA, Judge DP, Calkins H, Churko J, Wu JC, MacRae CA, Kleber AG, Saffitz JE. Identification of a new modulator of the intercalated disc in a zebrafish model of arrhythmogenic cardiomyopathy. Sci Transl Med. 2014 Jun 11;6(240):240ra74. doi: 10.1126/scitranslmed.3008008. PMID 24920660
- [Background] Chelko SP, Asimaki A, Andersen P, Bedja D, Amat-Alarcon N, DeMazumder D, Jasti R, MacRae CA, Leber R, Kleber AG, Saffitz JE, Judge DP. Central role for GSK3beta in the pathogenesis of arrhythmogenic cardiomyopathy. JCI Insight. 2016 Apr 21;1(5):e85923. doi: 10.1172/jci.insight.85923. PMID 27170944
- [Background] Roberts JD, Murphy NP, Hamilton RM, Lubbers ER, James CA, Kline CF, Gollob MH, Krahn AD, Sturm AC, Musa H, El-Refaey M, Koenig S, Aneq MA, Hoorntje ET, Graw SL, Davies RW, Rafiq MA, Koopmann TT, Aafaqi S, Fatah M, Chiasson DA, Taylor MR, Simmons SL, Han M, van Opbergen CJ, Wold LE, Sinagra G, Mittal K, Tichnell C, Murray B, Codima A, Nazer B, Nguyen DT, Marcus FI, Sobriera N, Lodder EM, van den Berg MP, Spears DA, Robinson JF, Ursell PC, Green AK, Skanes AC, Tang AS, Gardner MJ, Hegele RA, van Veen TA, Wilde AA, Healey JS, Janssen PM, Mestroni L, van Tintelen JP, Calkins H, Judge DP, Hund TJ, Scheinman MM, Mohler PJ. Ankyrin-B dysfunction predisposes to arrhythmogenic cardiomyopathy and is amenable to therapy. J Clin Invest. 2019 Jul 2;129(8):3171-3184. doi: 10.1172/JCI125538. eCollection 2019 Jul 2. PMID 31264976
- [Background] Padron-Barthe L, Villalba-Orero M, Gomez-Salinero JM, Dominguez F, Roman M, Larrasa-Alonso J, Ortiz-Sanchez P, Martinez F, Lopez-Olaneta M, Bonzon-Kulichenko E, Vazquez J, Marti-Gomez C, Santiago DJ, Prados B, Giovinazzo G, Gomez-Gaviro MV, Priori S, Garcia-Pavia P, Lara-Pezzi E. Severe Cardiac Dysfunction and Death Caused by Arrhythmogenic Right Ventricular Cardiomyopathy Type 5 Are Improved by Inhibition of Glycogen Synthase Kinase-3beta. Circulation. 2019 Oct;140(14):1188-1204. doi: 10.1161/CIRCULATIONAHA.119.040366. Epub 2019 Sep 5. PMID 31567019